CLINICAL TRIAL: NCT02968381
Title: A Guided Imagery Tobacco Cessation Intervention Delivered by a Quit Line and Website
Acronym: QLImagery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34AT008947 (NIH); 1R34AT008947 (NIH)
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Results first posted 2021-01-08 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Tobacco Use; Smoking Cessation; Smoking, Tobacco; Tobacco Smoking; Guided Imagery
Keywords: tobacco; smoking; imagery
MeSH Terms: conditions — Tobacco Use; Smoking Cessation; Tobacco Smoking; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery Intervention (Experimental): Participants will receive imagery intervention which includes 6 telephone sessions, an introduction to guided imagery, setting a quit date, setting guided imagery schedule, and a description of and instructions for using the study website.
  Interventions: Behavioral: Imagery Intervention
- Control Condition (Active Comparator): Participants will receive an attention control condition which includes 6 telephone sessions, an introduction to cognitive behavioral telephone coaching, setting a quit date, creating a quit plan, and a description of and instructions for using the Arizona Smokers' Help Line website.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Imagery Intervention — Telephone coaching sessions, use of guided imagery and website.
  Arms: Imagery Intervention
Behavioral: Control Condition — Telephone coaching using standard cognitive behavioral methods
  Other Names: Active Comparator
  Arms: Control Condition

SUMMARY:
Tobacco use is still the leading cause of preventable disease and death in the United States. Tobacco quit lines are effective at helping smokers to quit, but quit lines are underutilized, especially by men and racial/ethnic minorities. Guided imagery is effective at helping people quit smoking, and is appealing to males and diverse racial groups, but has limited reach. The proposed study will develop and test the feasibility and acceptability of a guided imagery tobacco cessation intervention that is delivered by a combination of quit line coaches and an interactive website. The investigators hypothesize that guided mental imagery delivered using the quit line "coaching model" combined with an interactive website could be an effective intervention strategy.

DETAILED DESCRIPTION:
The objective of this three year R34 application is to develop and test the feasibility of a theory-driven, telephone plus web-based, guided mental imagery intervention for smoking cessation.

Aim 1. Develop a theory-based, guided mental imagery tobacco cessation intervention for quit line callers with input from expert consultants in health disparities and a Community Advisory Board representing diverse populations and tobacco control stakeholders. The intervention will include phone-based coaching, an interactive website, and optional cessation medication. It will be focus tested with 40 smokers (from diverse racial/ethnic and age groups with at least 40% males), and usability tested with 5 smokers.

Aim 2. Develop training and competency standards for, and train, four coaches in the implementation of the guided imagery and control interventions. Coaches will be assessed at 6-weeks and 6-months post-training for implementation fidelity and satisfaction.

Aim 3. Conduct a feasibility trial (N=100) to gather preliminary data on the effects of the guided mental imagery intervention on quit line callers' tobacco use, cravings, and self-efficacy to quit smoking, and to refine study procedures, including recruitment, retention, and use of intervention components. Participants will be randomly assigned to receive either the Imagery Intervention (N=50) or an attention control condition (N=50) as delivered by study coaches. Participants will be assessed at baseline, 6-weeks and 6-months post-enrollment. Primary outcomes will be self-reported point prevalence and prolonged abstinence of tobacco use. Biochemical validation will be conducted on a sub-sample to determine validity of self-reported abstinence in this population. Secondary outcomes will be self-reported cravings and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker trying to quit
* Speak English
* Internet access
* Email access
* Live in the state of Arizona, USA

Exclusion Criteria:

* Having enrolled and participated in Quit line services in the past 12 months
* Diagnosed with a serious mental illness (e.g. current depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Gordon, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon JS, Bell ML, Armin JS, Giacobbi PR, Nair US. A telephone-based guided imagery tobacco cessation intervention: results of a randomized feasibility trial. Transl Behav Med. 2021 Mar 16;11(2):516-529. doi: 10.1093/tbm/ibaa052. PMID 32542352
- See also: Pilot project using guided imagery for tobacco cessation for women concerned about weight gain — http://SeeMeSmokeFree.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imagery Intervention | Control Condition
Started | 61 | 60
Completed | 56 | 50
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Population: Information on participants with available data is used in analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Imagery Intervention | Control Condition | Total
Number analyzed (Participants) | 56 | 49 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 48 | 104
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (15.8) | 51.6 (14.5) | 50.5 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 48 | 40 | 88
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 45 | 39 | 84
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 56 | 49 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Self-reported 7-day Tobacco Abstinence From Baseline to Follow-up
Description: Tobacco use over the past seven days is assessed by project staff at 6-months post-enrollment. Tobacco use includes cigarettes, smokeless tobacco, and other types of tobacco. The question is asked "Have you smoked, even a puff, in the last 7 days?" "Have you used any other form of tobacco in the last 7 days?" If yes to either question, the participant is asked to indicate what type of tobacco was used and how much was used (e.g., "how many cigarettes did you smoke on a typical day?").
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Imagery Intervention | Control Condition
Number analyzed (Participants) | 56 | 49
Participants | 15 | 21

2. Primary Outcome: Number of Participants With Change in Self-reported Tobacco 30-day Abstinence From Baseline to Follow-up
Description: Tobacco use over the past 30 days is assessed by project staff at 6-months post-enrollment. Tobacco use includes cigarettes, smokeless tobacco, and other types of tobacco. The question is asked "Have you smoked, even a puff, in the last 30 days?" "Have you used any other form of tobacco in the last 30 days?" If yes to either question, the participant is asked to indicate what type of tobacco was used and how much was used (e.g., "how many cigarettes did you smoke on a typical day?").
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Imagery Intervention | Control Condition
Number analyzed (Participants) | 56 | 49
Participants | 12 | 16

3. Secondary Outcome: Change in Tobacco Use for Non-quitters From Baseline to Follow-up
Description: Assessed by project staff at 6-months post-enrollment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Cigarettes
Arm/Group | Imagery Intervention | Control Condition
Number analyzed (Participants) | 56 | 49
Cigarettes | 9.1 (6.1) | 11.2 (9.0)

4. Secondary Outcome: Change in Self-efficacy for Quitting From Baseline to Follow-up
Description: An abbreviated version of the Condiotte and Lichtenstein (1981) Confidence Questionnaire consisting of 5 items for quitters and 6 items for non-quitters. All items are scored using a 5-point Likert scale where 1 is low/less and 5 is high/more. We calculated an average score of the items (which would have a value between 1 and 5).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Imagery Intervention | Control Condition
Number analyzed (Participants) | 56 | 49
units on a scale | 4.1 (1.1) | 4.0 (1.2)

5. Secondary Outcome: Change in Nicotine Cravings From Baseline to Follow-up
Description: This was assessed using 1 item adapted from the Shiffman (2004) Rating Scale ("How much have you craved tobacco today?"). Responses were coded using a 6-point Likert scale from "not at all" (code 0) to "a great deal" (code 5).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Imagery Intervention | Control Condition
Number analyzed (Participants) | 56 | 49
score on a scale | 2.1 (1.2) | 2.2 (1.7)

ADVERSE EVENTS:
Time Frame: 10 months
Description: The intervention and control conditions were both cognitive behavioral and posed no risk to participants.
Arm/Group | Imagery Intervention | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/49
Other Adverse Events (participants affected / at risk) | 0/56 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02968381/Prot_SAP_000.pdf